CLINICAL TRIAL: NCT03632447
Title: A Prospective Randomized Efficacy Study Comparing a Pelvic Digital Health System Home Program of Pelvic Floor Muscle Exercise to Kegel Exercises in the Treatment of Stress-Predominant Urinary Incontinence
Brief Title: Comparing Use of a Digital Health System of Pelvic Floor Exercise Program to Kegel Exercises in Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Renovia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REN-05
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2019-07

CONDITIONS: Stress Urinary Incontinence; Mixed Urinary Incontinence
Keywords: Digital Health; Female
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessments of pelvic floor muscle function accomplished by testing at baseline, 4-weeks (mid-study) and 8-weeks will be performed by blinded assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Leva Arm (Experimental): Subjects will undergo pelvic floor muscle training using the leva device (a vaginal probe) which provides immediate visual feedback via smartphone regarding the motion of pelvic floor muscles. Subjects will perform exercises 2 1/2 minutes twice daily for 8 weeks. At the beginning of the study, four weeks later, and eight weeks later subjects will undergo pelvic floor muscle testing using the PFDx device and surveys to document response to training. After eight weeks, subjects may pursue any additional treatments they wish, but may continue to use the device. They will be further randomized to receive reminder text messages or no messages over 10 months. Subjects will be asked to complete follow up surveys at 6- and 12-months.
  Interventions: Device: Leva; Device: PFDx
- Kegel Arm (Active Comparator): Subjects in this arm will perform pelvic floor muscle exercises (Kegels) for the treatment of stress or mixed urinary incontinence. Subjects will be asked to perform exercises three times daily for 8 weeks. At the beginning of the study, four weeks later, and eight weeks later, subjects will undergo pelvic floor muscle testing (using the PFDx device) and surveys to document response to training. After eight weeks, subjects may pursue any additional treatments they wish, but may continue to use the device.
  Interventions: Device: PFDx

INTERVENTIONS:
Device: Leva — Subjects randomized to Leva will use a vaginal probe containing motion-based sensors to direct the performance of pelvic muscle exercises.
  Arms: Leva Arm
Device: PFDx — All subjects (in both study arms) will be evaluated using a vaginally placed device that will evaluate pelvic floor motion to document change in pelvic floor muscle function resulting from pelvic floor muscle exercises.

SUMMARY:
A randomized controlled trial for patients with stress urinary incontinence or stress-dominant mixed incontinence. Subjects will be randomized to 8-weeks of home kegel exercises or 8 weeks of pelvic floor muscle exercises using the leva digital pelvic health system that includes visual biofeedback via smartphone.

DETAILED DESCRIPTION:
A randomized controlled trial for patients with stress urinary incontinence or stress-dominant mixed incontinence.Subjects will be randomized to 8-weeks of home kegel exercises or 8 weeks of pelvic floor muscle exercises using the leva digital pelvic health system that includes visual biofeedback via smartphone. Leva subjects will perform guided pelvic floor muscle exercises for 2 1/2 minutes twice daily. Home kegel subjects will perform kegel exercises three times daily. Following 8-weeks of training, subjects will be permitted to continue the exercises or pursue additional therapies as indicated. Subjects randomized to the leva digital health system will be further randomized to receive automated reminders for the remainder of one year, or no additional reminders.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent.
* Self-reported stress-type UI symptoms of >= three months duration
* Diagnosis of stress predominant urinary incontinence based on MESA stress symptom score greater than MESA urge symptom score (percent of total possible urge score).
* UDI-6 score >/= 25
* Willing to participate in the 8-week study with follow up at 6-and 12-months, refraining from the pursuit of treatment for Stress Urinary Incontinence using other modalities (i.e. will not wear a pessary, participate in pelvic floor PT or surgery) during the first 8- weeks.

Exclusion Criteria:

* Absence of a vagina.
* Age <18 years.
* Stage 3-4 pelvic organ prolapse (as determined by POP-Q).
* Diagnosis of any neuromuscular disease.
* Non-ambulatory.
* Currently pregnant or <12 months post-partum.
* </= 3 months after failed surgery for stress urinary incontinence.
* Previous pelvic floor muscle training (PFMT) within the last 12 months under a supervised therapeutic plan of care.
* Currently taking, or has taken within the last 2 months, medication to treat urinary incontinence.
* Prior augmentation cystoplasty or artificial sphincter.
* Implanted nerve stimulator for urinary symptoms.
* Participation in another clinical study within 30 days of screening.
* Impaired cognitive function.
* Contraindication to the use of a vaginal probe.
* Unable to understand instructions on the use of the leva® Plus Pelvic Digital Health System.
* Unable to actively recruit the pelvic floor muscles to any degree for attempted volitional contraction.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
PGI-I | 8 weeks after randomization
  PGI-I, Patient Global Impression of Improvement, is a five-point scale that ranges from "not at all" to "very much better."
UDI-6 | 8 weeks after randomization
  Urogenital Distress Inventory is a six question validated questionnaire evaluating incontinence symptoms. It is scored from 0-100, with higher scores indicating more severely bothersome symptoms

SECONDARY OUTCOMES:
3-day voiding diary | 8 weeks after randomization
  An objective evaluation of urinary incontinence

OTHER OUTCOMES:
Adherence | 8 weeks, 6 months, 12 months
  Adherence to the exercise regimen will be evaluated

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - Cedars-Sinai Medical Group, Beverly Hills, California
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - Univeristy of Oklahoma, Oklahoma City, Oklahoma
  - Urology San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT03632447/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT03632447/SAP_002.pdf